CLINICAL TRIAL: NCT03415698
Title: Granulocyte Colony Stimulating Factor in Decompensated Cirrhosis: an Open Label Study
Brief Title: G-CSF in Decompensated Cirrhosis: an Open Label Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCSF in cirrhosis
Record Dates: First submitted 2018-01-11; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Cirrhosis, Liver
Keywords: Regenerative medicine
MeSH Terms: conditions — Liver Cirrhosis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Therapy (Active Comparator): Standard medical therapy will include nutritional support, rifaximin, lactulose, bowel wash, albumin, diuretics, multivitamins, antibiotics. fresh frozen plasma and packed red-cell transfusions (as required)
  Interventions: Drug: Standard Medical Therapy
- G-CSF + Standard Medical Therapy (Active Comparator): G-CSF at the dosage of 5 µg/Kg subcutaneously every 12 hr will be administered for five consecutive days. Four such cycles at 3 monthly intervals will be administered.
  Interventions: Drug: G-CSF; Drug: Standard Medical Therapy

INTERVENTIONS:
Drug: G-CSF — G-CSF will be administered at the dosage of 5 µg/Kg subcutaneously every 12 hr for five consecutive days. four such cycles will be administered at three monthly intervals.
  Arms: G-CSF + Standard Medical Therapy
Drug: Standard Medical Therapy — Nutritional support, rifaximin, lactulose, bowel wash, albumin, diuretics, multivitamins and antibiotics.

SUMMARY:
Globally, cirrhosis is the fifth commonest cause of mortality. Its natural history is typified by an initial, largely asymptomatic, "compensated" phase followed by "decompensation" due to complications of raised portal pressures and hepatocellular dysfunction.

Currently the only definitive treatment option for cirrhosis is liver transplantation which is limited in its applicability due to donor shortage, exorbitant costs and lack of widespread availability. The need for long term immunosuppression and its attendant complications are a further drawback. The ability of stem cells to differentiate into multiple cellular lineages makes one speculate that they can be used for tissue repair and regeneration when tissue-resident stem cells become overwhelmed. Bone marrow derived stem cells have amazing plasticity. They can "home" to the liver in response to injury and help in liver regeneration by trans-differentiation, cell fusion and augmentation of tissue- resident stem cell mediated repair. Two methods are available for the mobilisation of stem cells from the bone marrow to the liver. One involves the administration of cytokines like granulocyte-colony stimulating factor (G-CSF) and the other is the isolation of stem cells from the marrow followed by their injection into the hepatic artery or portal vein after purification. The latter is probably more cumbersome and may be potentially risky due to the underlying coagulation abnormalities in cirrhotic patients .

G-CSF has been shown to mobilise bone marrow stem cells and even increase survival in patients of severe alcoholic steatohepatitis and ACLF. There is conflicting evidence on the role of G-CSF in decompensated cirrhosis with some studies showing improved survival while others have shown a lack of clinical or biochemical benefit. Many of these studies have used a single course of G-CSF. Verma et al, in a recent study published in 2018, elegantly demonstrated the beneficial effect of multiple courses of G-CSF in improving mortality and transplant free survival in decompensated cirrhotics.

The investigators too speculate that multiple cycles of G-CSF could result in better outcomes in decompensated cirrhosis by causing more prolonged and sustained stem cell homing to the liver. Thus, this study is being undertaken to further evaluate the safety and efficacy of multiple cycles of G-CSF in decompensated cirrhotics.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated Cirrhosis of liver irrespective of etiology

Exclusion Criteria:

* Acute on chronic liver failure (fulfilling either APASL or CANONIC criteria of ACLF)
* Splenic diameter of more than 18 cm
* Concomitant HCC or other active malignancy
* Upper gastrointestinal bleeding in the previous 7 days
* Portal vein thrombosis
* Severe renal dysfunction as defined by creatnine > 1.5mg/dl
* Severe cardiac dysfunction
* Uncontrolled diabetes (Hb A 1c ≥ 9) or diabetic retinopathy
* Acute infection or disseminate intravascular coagulation
* Active alcohol abuse in last 3 months
* Known hypersensitivity to G-CSF
* HIV co-infection
* Pregnancy
* Refusal to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Survival | One year
  Survival at 1 year after start of therapy

SECONDARY OUTCOMES:
Hemopoieticstem cell mobilisation | One Year
  Mobilisation of CD 34+ cells in peripheral blood
Clinical improvement in liver functions | One Year
  Occurrence of decompensations namely ascites, hepatic encephalopathy and variceal bleed
Biochemical improvement in liver functions | One year
  Improvment in MELD score
Improvement in nutritional status | One Year
  Nutritional status will be assesses by skeletal muscle index measurement using CT scan measurements at L3 level
Improvement in quality of life | One year
  Quality of life will be assessed using SF-36V2 Health Survey questionnaire
Safety of G-CSF as assessed by its adverse effects | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, DM, Principal Investigator — Professor, Department of Hepatology, PGIMER, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaur A, Verma N, Singh B, Kumar A, Kumari S, De A, Sharma RR, Singh V. Quantitative liver SPECT/CT is a novel tool to assess liver function, prognosis, and response to treatment in cirrhosis. Front Med (Lausanne). 2023 Mar 22;10:1118531. doi: 10.3389/fmed.2023.1118531. eCollection 2023. PMID 37035316
- [Derived] De A, Kumari S, Singh A, Kaur A, Sharma R, Bhalla A, Sharma N, Kalra N, Singh V. Multiple Cycles of Granulocyte Colony-Stimulating Factor Increase Survival Times of Patients With Decompensated Cirrhosis in a Randomized Trial. Clin Gastroenterol Hepatol. 2021 Feb;19(2):375-383.e5. doi: 10.1016/j.cgh.2020.02.022. Epub 2020 Feb 21. PMID 32088302